CLINICAL TRIAL: NCT05897112
Title: Comparison of 10% Potassium Hydroxide Solution Versus Cryotherapy in the Treatment of Molluscum Contagiosum
Brief Title: Comparative Efficacy of 10% Potassium Hydroxide Solution Versus Cryotherapy in Molluscum Contagiosum
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Combined Military Hospital Abbottabad (Other)
Responsible Party: Principal Investigator, danyal sajjad, Principal Investigator, Combined Military Hospital Abbottabad
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CMHAbbottabad22
Record Dates: First submitted 2023-05-19; First posted 2023-06-09 (Actual); Last update posted 2023-06-09 (Actual); Status verified 2023-05

CONDITIONS: Molluscum Contagiosum
MeSH Terms: conditions — Molluscum Contagiosum

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A received cryotherapy (Active Comparator): Group A were subjected to weekly cryotherapy with a cotton stick dip ped in Liquid Nitrogen for 02 Freezes and Thaw Cycle of 07 seconds with each cycle 10 seconds apart for 3 weeks
  Interventions: Drug: Group A received cryotherpay
- Group B received 10% Potassium Hydroxide Solution (Active Comparator): Group B applied 10% Potassium Hydroxide solution twice daily with the help of a cotton tip applicator until lesion showed signs of inflammation or clearance for 3 weeks
  Interventions: Drug: Group B received 10% Potassium Hydroxide Solution

INTERVENTIONS:
Drug: Group A received cryotherpay — Group A were subjected to weekly cryotherapy with a cotton stick dip ped in Liquid Nitrogen for 02 Freezes and Thaw Cycle of 07 seconds with each cycle 10 seconds apart for 3 weeks
  Arms: Group A received cryotherapy
Drug: Group B received 10% Potassium Hydroxide Solution — Group B applied 10% potassium hydroxide aqueous solution twice daily with the help of a cotton tip applicator until lesion showed signs of inflammation or clearance for 3 weeks
  Arms: Group B received 10% Potassium Hydroxide Solution

SUMMARY:
A total of sixty patients presented to the outpatient dermatology department of Combined military hospital (CMH) Abbottabad with signs of molluscum contagiosum clinically diagnosed meeting inclusion criteria were enrolled. Sample size was calculated using WHO sample size calculator. They were divided into two groups i.e Group A and Group B using lottery method. Patients in Group A were subjected to cryotherapy (liquid nitrogen gas) whereas patients in Group B patients were subjected to 10% potassium hydroxide solution for 3 weeks and were followed up at 2nd, 4th, 8th and 12th week for observing the progress of therapy in both groups on each follow up visit and ascertaining the efficacy respectively.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of molluscum contagiosum having 3-20 lesion
* no history of treatment before
* willingness to participate (given by parents)

Exclusion Criteria:

* Patients with facial lesions
* known immunodeficiency
* tendency for hypertrophic scarring
* known hypersensitivity

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Efficacy was assessed at 12th week by the clearance of lesion or not | 12 weeks
  Final evaluation in terms of efficacy was done at the follow up visit in 12th week and the method was termed as effective (Yes) on achieving complete clearance of lesions confirmed on clinical & physical examination of the affected areas by a consultant dermatologist using dermoscopy showing complete resolution of lesions. However, if lesions were not completely cleared at the end of 12th week, the treatment method was labelled as ineffective (No).

CONTACTS AND LOCATIONS:
Locations (1):
- CMH Abbottabad, Abbottābād, Khyber Pakhtunkhwa, Pakistan